CLINICAL TRIAL: NCT05093153
Title: Spanish Registry of Patients With Diagnosis of IgM-MGUS, Asymptomatic & Symptomatic Waldenström Macroglobulinemia. Analysis of Clinical and Laboratory Features, Treatment and Outcomes.
Brief Title: Spanish Registry of Patients With IgM Monoclonal Gammopathies
Acronym: PRAME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Española de Hematología y Hemoterapía (Other)
Responsible Party: Sponsor
Other Study IDs: PRAME
Record Dates: First submitted 2021-09-28; First posted 2021-10-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-11

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Waldenström's macroglobulinemia cohort patient: Adult patients diagnosed with Waldenström's Macroglobulinemia

SUMMARY:
Waldenström's macroglobulinemia (WM) is a B-cell lymphoproliferative disorder which is defined by bone marrow infiltration by small lymphocytes, lymphoplasmacytoid and plasma cells together with the presence of a detectable monoclonal immunoglobulin M (IgM).The clinical presentation of WM is variable. Symptoms can be related to tumor infiltration, or they can be related to the monoclonal IgM component. The therapeutic options are heterogeneous and there are no well-established in both first line or relapse/refractory settings. In Spain, the incidence of MGUS-IgM and WM in the last decade is unknown.

The aims of this retrospective, observational, multicentric study is:

* To develop a national registry of patients diagnosed with Waldenström's Macroglobulinemia and Monoclonal Gammopathy of uncertain significance -IgM in Spain in the past 30years.
* To evaluate the most relevant clinical characteristics, long-term safety and efficacy of different therapeutic schemes and long-term prognosis of patients with WM
* To help in the design of future therapeutic strategies, risk prognostic factors and clinical trials in Spain.

Methods:

The investigators will collect data from the patient clinical files after prior Informed Consent providing from patients with diagnosis of MGUS-IgM and WM in the past 30 years in Spain, according to the WHO classification of lymphoid tumors (2008) revised in 2016. Data from patients not able to provide IC (i.e., already dead patients) will be included only after the permission of the ethics review board.

The collected data will be included in a database of the Spanish Myeloma and Lymphoma Intergroup (SMALI) team created ad-hoc by the Spanish Society of Hematology and Hemotherapy (SEHH). Each principal investigator in each center will conduct their technical supervision. The evaluation of the treatment protocols will be done following the indications of the intergroup committee according to the guidelines of the International Waldenström's Macroglobulinemia Group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients having a confirmed diagnosis of either in the las 30 years:
* Monoclonal Gammopathy of uncertain significance -IgM
* Asymptomatic Waldenström's macroglobulinemia
* Symptomatic Waldenström's macroglobulinemia

Exclusion Criteria:

* Other subtypes of Lymphoproliferative diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Waldenström's Macroglobulinemia and Monoclonal Gammopathy of uncertain significance
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 4 years
  Overall survival evaluation from the date of diagnosis to the death of the patient due to any cause

CONTACTS AND LOCATIONS:
Locations (32):
- Spain (32):
  - Hospital Son Llatzer, Palma, Balearic Islands
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - ICO Badalona - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Déu de Manresa, Manresa, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - CUN Navarra, Pamplona, Navarre
  - Hospital Vital Álvarez-Buylla, Mieres, Principality of Asturias
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Complejo Hospitalario Universitario de La Coruña (CHUAC), A Coruña
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Clínico San Cecilio, Granada
  - CAU de León, León
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Universitario Fundación Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - CAU de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Clínico de Valencia, Valencia
  - Hospital La Fe de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No